CLINICAL TRIAL: NCT05090332
Title: Effects of Dry Needling Versus Fascial Gun on Pain Pressure Threshold, Cervical Ranges in Patients With Active Trigger Points of Trapezius Muscle.
Brief Title: Comparison of Dry Needling and Thera Gun Treatment on Trapezius Muscle Active Trigger Points.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01062 Dr Hira Naz
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Neck Pain
Keywords: Trapezius Trigger Points; Range of motion; Pain threshold; Thera Gun; Dry Needling
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial Gun (Experimental): Vibrations through Facial gun along with conventional Therapy
  Interventions: Other: Facial Gun; Other: Dry Needling
- Dry needling (Experimental): Dry needling along with conventional treatment.
  Interventions: Other: Facial Gun; Other: Dry Needling

INTERVENTIONS:
Other: Facial Gun — Vibration massage applied for five Minutes directly on the trigger point
Other: Dry Needling — For dry needling the outer skin should be clean with alcohol and the taut band should be placed between thumb and index finger. Without damaging any nerve or artery the needle is passed though the muscle into the trigger point and breaking it to relief pain

SUMMARY:
Comparison of dry needling and Thera Gun on treatment of Active trigger points of trapezius Muscle, pain threshold and Range of motion of neck.

DETAILED DESCRIPTION:
Chronic neck pain related to the myo-facial systems from local muscle fiber contractions referred to "myo-facial trigger points" (MTrPs).MTrPs are highly sensitive spots that lie in the skeletal muscle, and are diagnosed with mechanical pressure, they can also develop as referral pain in a specific pattern. Although MTrPs are found in all muscle groups, they are more prevalent in the upper quarter postural muscles, especially the upper trapezius muscle.

Data will be collected from both gender patients having active trigger points in trapezius muscles. Then patients will be divided randomly into two groups. All patient will be given conventional treatment and then group A will be given treatment with Thera Gun and group B will be given dry needling treatment and then will compare effects of both.

To date, a wide range of physical therapy interventions have been suggested to address MTrPs including manual therapies (massage, stretching, myofascial release), electrotherapy modalities (surface heat, ultrasound, Transcutaneous Electrical Nerve Stimulator and laser therapy) and invasive techniques such as dry needling (DN) but none of study is done on the effectiveness of facial gun in decreasing pain intensity and increasing range of motion and none of study compare the effect of Dry needling with facial gun. So, this study will determine the effect of facial gun on pain intensity and range of motion and compare that effect with dry needling.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical pain due to active trigger points of trapezius muscle
* Numeric Pain Rating Scale> 3

Exclusion Criteria:

* Any previous history of Trauma or surgery
* Spondylitis
* Carcinoma
* Tuberculosis of spine
* Diagnosed with cervical pain & stiffness due to disc herniation, radiculopathy or any other cervical malignancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Three weeks
  Visual analogue scale (VAS) very simple and often used method to measure the intensity of pain or the attitude of the individual that may not be measured directly through any test. This scale has high degree of sensitivity i.e a discriminating capacity higher than the other scales. It is the continuous scale for estimation of the extent of pain consist of the straight line shows two extreme ends one is zero pain and the other is extreme pain and in between the words on far extreme 'slight, moderate and severe' too that is experience by the individual. When the patient fills the Visual analogue scale, the patient may mark the level of pain he/she experienced by highlighting the exact level along the line between these two ends. Assessment to be done at baseline, 3rd visit and 9th visit
Goniometer for cervical range of motion | Three weeks
  Goniometer is the instrument that measures the available range of the motion of joint. The goniometer is simple 360 degree with fulcrum and two arms. There are many types of goniometer one of them is universal standard goniometer that is consist of one moveable arm and the other is static (immobile) arm. That is either made of plastic or metal tool. It may help to measure the ranges of motions and their lengths. Inter-rater reliability (ICC2,2 = 0.79-0.92). Assessment to be done at baseline, 3rd visit and 9th visit
Algometer | Three weeks
  The pressure algometer (PA) is a measuring instrument that may help in the calculation of pain threshold for the involved trigger point. The force recorded is the amount of the pressure that caused pain in the subject called the pressure pain threshold. The inter-examiner reliability if the PA is good or satisfactory with the interclass correlation coefficient (ICC 0.78-0.93) . Assessment will be done at baseline, 3rd and 9th visit.

SECONDARY OUTCOMES:
Neck Disability Index | Three weeks
  Neck disability index: it is the assessment tool used for both research and clinical purposes for the measurement of chronic neck pain. The patient is asked to fill the questionnaire by the researcher or clinician in order to know the level of pain while managing its affects in daily life. Basically, the questionnaire is designed to assess the Activities of Daily livings and Instrumental Activities of daily Livings of patient complaining about chronic neck pain. There are 10 questions includes, pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each question is marked on a 0 to 5 rating scale where 0 is considered as 'no pain' and 5 means 'maximum pain'. Assessment to be done at baseline, 3rd and 9th visit.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, DSc PT, Principal Investigator — Riphah International University
Locations (1):
- Federal Government Polyclinic Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No